CLINICAL TRIAL: NCT00705107
Title: Evaluation of Adherence Rate in Patients Receiving PegIntron Pen / Rebetol for Hepatitis C
Brief Title: Adherence to Treatment With PegIntron Pen Plus Rebetol in Treatment-naïve Adult Patients With Hepatitis C in Romania (Study P04247)
Status: Terminated | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04247
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Treated Patients: All patients participating in the study
  Interventions: Biological: PegIntron pen (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron pen (peginterferon alfa-2b; SCH 54031) — PegIntron administered in accordance with approved labeling.
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered in accordance with approved labeling
  Other Names: SCH 18908

SUMMARY:
Adherence to the prescribed treatment regimen with PegIntron and Rebetol affects the chance of achieving a sustained virologic response in patients with hepatitis C. The objective of this study is to evaluate the proportion of patients who complete treatment with PegIntron pen and Rebetol while participating in a patient assistance program. The patient assistance program can consist of prophylactic treatment (eg, with growth factors, psychiatric medications) or other interventions (eg, psychotherapy, patient support groups, visiting nurse, nurse telephone calls, educational literature).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve patients with hepatitis C
* Patients treated with PegIntron pen and Rebetol
* Patients receiving patient assistance program

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment-naïve adult patients with hepatitis C treated with PegIntron pen and Rebetol receiving a patient assistance program at approximately 40 sites in Romania. Patient assistance program can consist of prophylactic treatment (eg, with growth factors, psychiatric medications) or other interventions (eg, psychotherapy, patient support groups, visiting nurse, nurse telephone calls, educational literature).
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2004-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Treated Patients
Started | 267
Completed | 218
Not Completed | 49

BASELINE CHARACTERISTICS:
Arm/Group | All Treated Patients
Number analyzed (Participants) | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.35 (10.11)
Sex/Gender, Customized [Number; unit: participants]
  Female | 168
  Male | 98
  Missing | 1
Region of Enrollment [Number; unit: participants]
  Romania | 267

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Completed Treatment.
Time Frame: Assessed at the end of the 48-week treatment.
Population: All participants
Measure: Number; unit: Participants
Arm/Group | All Treated Patients
Number analyzed (Participants) | 267
Participants | 218

2. Secondary Outcome: Average Length of Treatment.
Time Frame: Assessed at the end of treatment. The prescribed treatment duration was 48 weeks.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | All Treated Patients
Number analyzed (Participants) | 267
weeks | 43.60 (21.38)

ADVERSE EVENTS:
Arm/Group | All Treated Patients
Serious Adverse Events (participants affected / at risk) | 1/267
Other Adverse Events (participants affected / at risk) | 124/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=267)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Patients (N=267)
Anaemia (Blood and lymphatic system disorders) | 52 (148)
Leukopenia (Blood and lymphatic system disorders) | 28 (85)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (49)
Asthenia (General disorders) | 58 (163)
Chills (General disorders) | 15 (22)
Influenza like illness (General disorders) | 25 (62)
Pyrexia (General disorders) | 33 (60)
Weight decreased (Investigations) | 51 (86)
Decreased appetite (Metabolism and nutrition disorders) | 29 (68)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (30)
Headache (Nervous system disorders) | 25 (57)
Depression (Psychiatric disorders) | 18 (44)
Insomnia (Nervous system disorders) | 20 (48)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No